CLINICAL TRIAL: NCT05260567
Title: A Multimodal Tele-health Behavioural Intervention in Patients With Peripheral Arterial Disease From Low Socio-economic Areas: a Feasibility and Pilot Randomized Controlled Trial With Embedded Process Evaluation
Brief Title: Telehealth Exercise Training in Peripheral Arterial Disease - TEXT-PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Gabriel Cucato, Vice Chancellor Research Fellow, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 286735
Record Dates: First submitted 2022-02-15; First posted 2022-03-02 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication; Behavior, Health; Exercise Intervention
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Health Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and Lifestyle Change (Experimental): Exercise training and lifestyle change
  Interventions: Behavioral: Exercise and Lifestyle Change
- Standard Care (Other): Patients will also receive specific advice to perform an unsupervised walking exercise according to NICE guideline.
  Interventions: Behavioral: Exercise and Lifestyle Change

INTERVENTIONS:
Behavioral: Exercise and Lifestyle Change — Patients will undergo to weekly phone call/videoconference for 12 weeks and discuss the behaviour change.
  They also will undergo to home-based exercise training will be performed twice a week for 12 weeks via Zoom (up to 5 patients per session). Each session will be comprised of warm-up (10 min), the main part (15 to 20 min), and cooldown (5 to 10 min). The training aims to develop resistance, aerobic and functional capacity such as getting up, walking, pulling, pushing, throwing, transferring body weight or external loads. In addition, patients will be encouraged to increase their physical activity. Patients will be provided with a Fitbit device to monitor their step count and will be recommended to increase their previous week's average step count by 10%.

SUMMARY:
Peripheral arterial disease is a common, under-treated and under-researched issue. The vast majority of these patients often have multiple issues which can be improved with targeted behavioural change interventions. NICE has recommended that supervised exercise is the mainstay of treatment for intermittent claudication (ischaemic muscle pain on walking due to blocked and narrowed arteries). However, in the vast majority of UK hospitals, this isn't undertaken, and with the issues around group-based sessions and repeated visits to hospitals, this treatment option is not available with the coronavirus pandemic.

This is a single-centre randomised control trial in 60 patients with peripheral arterial disease attending the Freeman Hospital. Patients will be randomised to either an enhanced behavioural change intervention targeting multiple health behaviours vs a simple walking intervention. Also, some patients will be involved in focus groups to understand their experience of the intervention and whether it is feasible and acceptable, allowing changes to be made to the program.

The primary outcome will be to assess the feasibility and acceptability of the program. We will also be assessing multiple secondary outcomes including functional capacity, quality of life, sleep quality and smoking and alcohol reduction.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PAD confirmed by ankle-brachial index <0.90 in one or both limbs
* Age >= 40 years
* Able to walk distance >50m
* Live in an area deemed in lowest 30% of super output area from Office of National Statistics

Exclusion Criteria:

* chronic limb threatening ischemia
* short claudication distance <50m
* severe heart disease (Grade III or IV, New York Heart Association)
* severe ischemic or haemorrhagic stroke or neurodegenerative diseases
* severe hypertension (systolic blood pressure of more than 180 mm Hg, and a diastolic
* blood pressure of more than 100 mm Hg)
* uncontrolled cardiac arrhythmias (unstable angina during the previous month and
* myocardial infarction during the previous month)
* a resting heart rate of more than 120 beats per minute
* has already undergone angioplasty, bypass or other surgical intervention for PAD
* other severe comorbid conditions preventing the ability to engage in physical activity,
* inability or unwillingness to undertake the commitments of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-05 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of the program | post 12 weeks
  Feasibility will be determined by calculating the rate of patient screening, eligibility, recruitment, retention at 12 weeks and adherence to the intervention (number of sessions attended and completed)
Acceptability of the program | post 12 weeks
  Patient acceptability of the intervention and study experience more broadly will be determined through semi-structured qualitative 1-2-1 interviews and/or focus groups.

SECONDARY OUTCOMES:
Six-minute walk test (6MWT) | pre and post-12 weeks
Walking Impairment Questionnaire (WIQ) | pre and post-12 weeks
Walking Estimated Limitation Calculated by History (WELCH) questionnaire | pre and post-12 weeks
Vascular quality of life questionnaire (VascuQoL-6) | pre and post-12 weeks
EuroQoL questionnaire (EQ-5D-5L). | pre and post-12 weeks
Short Form Dietary Questionnaire | pre and post-12 weeks
Physical activity levels (Fitbit Charge HR) | pre and post-12 weeks
Sleep | pre and post-12 weeks
  (Fitbit Charge HR)
Alcohol and tobacco use | pre and post-12 weeks
  The 3-item Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) and self-reported smoking habits
Mental wellbeing | pre and post-12 weeks
  hospital anxiety-depression score (HADS)
Patient activation | pre and post-12 weeks
  The Patient Activation Measure (PAM®)
Resource utilisation | pre and post-12 weeks
  The case report forms (CRF)

CONTACTS AND LOCATIONS:
Overall Officials: James Prentis, Principal Investigator — Freeman Hospital - Newcastle upon Tyne NHS trust
Locations (1):
- Freeman Hospital - Newcastle upon Tyne NHS trust, Newcastle upon Tyne, United Kingdom